CLINICAL TRIAL: NCT04665674
Title: Enquête épidémiologique Sur la prévalence et le Pronostic de l'Histiocytose Langerhansienne Pulmonaire de l'Adulte en France
Brief Title: Adult Pulmonary Langerhans Cell Histiocytosis: a National Registry-based Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2014_TAZI
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Histiocytosis; Histiocytosis, Langerhans-Cell; Histiocytosis Pulmonary
MeSH Terms: conditions — Histiocytosis; Histiocytosis, Langerhans-Cell | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Langerhans cell histiocytosis (PLCH): All patients with newly diagnosed PLCH at adulthood (i.e. 18 years of age or older) referred to the French national reference centre for Histiocytoses
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Standard of car of pulmonary Langerhans cell histiocytosis (PLCH)

SUMMARY:
The long-term outcomes of adult patients with pulmonary Langerhans cell histiocytosis (PLCH), particularly survival, is largely unknown. This is the first prospective study in the field evaluating the long-term outcomes of PLCH patients. This french countrywide registry-based study included a large cohort of PLCH patients followed for a sufficiently long period to address risk factors of long-term outcomes of PLCH patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of PLCH was either histologically confirmed on a biopsy of an involved tissue, or based on the combination of the following criteria: 1) an appropriate clinical picture; 2) a typical nodulo-cystic pattern on lung high-resolution computed tomography (HRCT) and 3) exclusion of alternative diagnoses

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with newly diagnosed PLCH at adulthood (i.e. 18 years of age or older) referred to the French national reference centre for Histiocytoses
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 20 years
  Overall survival defined as the time from inclusion to death from any cause.

SECONDARY OUTCOMES:
CRF | 20 years
  Cumulative incidence of chronic respiratory failure (CRF) from inclusion
PH | 20 years
  Cumulative incidence of pulmonary hypertension (PH) from inclusion
Malignant diseases | 20 years
  Cumulative incidence of Malignant diseases from inclusion
Extra-pulmonary involvement in isolated PLCH | 20 years
  Cumulative incidence of extra pulmonary localisations from inclusion
Annual prevalence | 20 years
  Number of people with the disease at any time during a year

CONTACTS AND LOCATIONS:
Locations (1):
- French national reference centre for Histiocytoses, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benattia A, Bugnet E, Walter-Petrich A, de Margerie-Mellon C, Meignin V, Seguin-Givelet A, Lorillon G, Chevret S, Tazi A. Long-term outcomes of adult pulmonary Langerhans cell histiocytosis: a prospective cohort. Eur Respir J. 2022 May 26;59(5):2101017. doi: 10.1183/13993003.01017-2021. Print 2022 May. PMID 34675043